CLINICAL TRIAL: NCT03167996
Title: Chronic Cardiovascular Risk Outpatient Management in South Asians Using Digital Health Technology
Acronym: HealthPals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: HealthPals, Inc (Unknown)
Responsible Party: Principal Investigator, Shriram Nallamshetty, Clinical Assistant Professor (Affiliated) [VAPAHCS], Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 36464
Record Dates: First submitted 2017-05-15; First posted 2017-05-30 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Cardiovascular Risk Factor; Insulin Resistance; PreDiabetes; Diabetes; Coronary Artery Disease; Hypertension; Prehypertension; Dyslipidemias
Keywords: South Asian; Cardiovascular Risk Reduction; Metabolic Disorders; Lifestyle modifications
MeSH Terms: conditions — Insulin Resistance; Prediabetic State; Diabetes Mellitus; Coronary Artery Disease; Hypertension; Prehypertension; Dyslipidemias; Metabolic Diseases

STUDY DESIGN:
Intervention Model Description: Group A Control Group B HealthPals
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group B/ HealthPals (Experimental): Group B have access to HealthPals app where they will coordinate with a trained health coach Group B patients will only come into SSATHI clinic to see their doctor for an initial visit and 6 month follow up, and they will have a telephone visit with their doctor at 3 months instead of an in-clinic visit
  Lab testing is the same for both Group A/ control and Group B patients
  Interventions: Behavioral: Use of HealthPals (Telemedicine supported by digital health platform)
- Group A/ Control (No Intervention): Group B will not have access to HealthPals app
  Group A patients will come into SSATHI clinic to see their doctor for an initial visit, a 3 month follow up, and a 6 month follow up
  Lab testing is the same for both Group A/ control and Group B patients

INTERVENTIONS:
Behavioral: Use of HealthPals (Telemedicine supported by digital health platform) — HealthPals is a smartphone-based chronic disease management mobile application. It uses the mobile health capabilities of smartphones to provide a secure communication portal for patients with their Care Teams to help achieve cardiovascular risk reduction through a digital health coach-based coaching for lifestyle and medication compliance.
  The HealthPals app was developed by HealthPals, Inc.
  Arms: Group B/ HealthPals

SUMMARY:
This platform will enable investigation the cardiovascular risk reduction and the increase in participant engagement in their heart-healthy goals, through the use of virtual care/telemedicine with a digital platform that connects them to their own doctors, nurses, and dietitians.

DETAILED DESCRIPTION:
The study will use telemedicine and the mobile health capabilities of smartphones to facilitate communication of medical goals set by the treating physician to the subject in between clinic visits, and to assess the daily medical and lifestyle change compliance of enrolled Stanford subjects and provide virtual health coaching, as needed, to subjects to achieve said goals. How patients comply with their specific medical and lifestyle goals all affect their cardiovascular health, yet largely go unmeasured. These can now be measured with a notification-based system in which subject-entered activity, medication compliance, and dietary reporting data will be collected, assessed, and trigger appropriate responses by the subject's Care Team, which includes their physician, nurse, dietitian, and assigned health coach. We aim to collect this subject-reported activity and cardiovascular care plan compliance data to provide much more quantitative data on type, duration, and intensity of daily activities and compliance with the medication regimens of enrolled subjects.

The study will compare anthropometric cardiovascular risk biomarkers testing at the initial visit and after 3 months, in subjects utilizing the HealthPals digital platform PLUS the standard SSATHI clinic visits, versus subjects receiving only SSATHI clinic visits.

ELIGIBILITY:
Inclusion Criteria:

* adult smartphone users

Exclusion Criteria:

* Subjects who do not own a smartphone or cannot access their mobile health data
* Patients unable to read English, as the initial version of the research app will be in English
* Participants who are children (under 18 years old)
* Participants who are pregnant women
* Participants who are economically and educationally disadvantaged, decisionally impaired, homeless people, or employees of Stanford University will be excluded due to being of a vulnerable population.
* Participants who express active chest pain or shortness of breath in their first clinic visit and are clinically deemed to require an emergency room evaluation will be excluded
* Participants who have inability or unwillingness to use or connect to data services for app messaging
* Participants with an upcoming surgical procedure (for instance, a clinic visit as part of preoperative evaluation) that will significantly impair or block their ability to follow the chronic disease management program during the study period
* Participants who have pre-existing participation in another clinical research protocol.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2016-06-23 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-03-23 (Actual)

PRIMARY OUTCOMES:
Change in exercise activity over 6 months | 6 months or through study completion
  Patients are given exercise recommendations (or physical activity goals depending on the patient's capacity for exercise) at the time of the initial visit by the HealthPals health coach. The patients will input their activity into the HealthPals platform at time points of their convenience during their 6 month involvement in the study, and this data will be securely aggregated within the platform. The HealthPals health coach who has access to this data will compile and analyze the data and also send it back to the patients' providers by means of final health reports, assessing the change of exercise activity over the duration of the patient's involvement in the study.
Measuring medication compliance | Monthly assessment and report for duration of their involvement in the study
  The patients will input their compliance to their medication regimen into the HealthPals platform at time points of their convenience, and this data will be securely aggregated within the platform. The HealthPals health coach who has access to this data will compile and analyze the data and also send it back to the patients' providers by means of final reports.
Measuring trends in Blood Pressure measurements | Monthly assessment and report for duration of their involvement in the study
  The patients will input their blood pressure in mmHg at time points of their convenience into the HealthPals platform, and this data will be securely aggregated within the platform. The HealthPals health coach who has access to this data will compile and analyze the data and also send it back to the patients' providers by means of monthly health reports.
Measuring trends in weight measurements | Monthly assessment and report for duration of their involvement in the study
  The patients will input their weight in kg at time points of their convenience into the HealthPals platform, and this data will be securely aggregated within the platform. The HealthPals health coach who has access to this data will compile and analyze the data and also send it back to the patients' providers by means of monthly health reports.
Measuring compliance to dietary recommendations | Monthly assessment and report for duration of their involvement in the study
  Patients are given dietary recommendations at the time of their initial visit by the HealthPals health coach. After the first visit the patients will input their diet into the HealthPals platform at time points of their convenience, and this data will be securely aggregated within the platform. The HealthPals health coach who has access to this data will compile and analyze the data and also send it back to the patients' providers by means of monthly health reports.
Initial User Assessment | Questionnaire administered at time of initial visit
  Questionnaire covering personal history, family history, typical diet, exercise and activity, and stress level quantification. This questionnaire is used for a baseline analysis of the patients' health status by the HealthPals health coach.

CONTACTS AND LOCATIONS:
Overall Officials: Fahim Abbasi, MD, Principal Investigator — Stanford University; Shriram Nallamshetty, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No